CLINICAL TRIAL: NCT04889482
Title: Functional Testing and Performance in Tennis
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Principal Investigator, University of Liege
Other Study IDs: Functional testing tennis
Record Dates: First submitted 2020-03-09; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Tennis
Keywords: tennis serve, performance, functional testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study was to correlate functional tests, clinical tests and rotator cuff strength with the speed of serve.

For that purpose, tennis players (ITN 2-4) will be recruted among tennis players in the Province of Liege. They will be assessed 2 times.

During the first assessment, lateral medicine ball throw, 2 ball throws, upper extremity y balance test and shoulder rotation range of motion will be assessed.

During the second assessment, lateral medicine ball throw, the 2 ball throws and rotator cuff strength will be assessed.

DETAILED DESCRIPTION:
Forty healthy tennis players (ITN 2-4) will be recruted among players in the club of the Province of Liege.

First session :

* Clinical testing

  1. Upper extremity Y Balance Test
  2. Range of motion (internal/external rotation)
* Functional tests

  a. Lateral Medecine Ball throw (5 repetitions) b. Single arm ball throw (1,5kg) d. Core endurance test
* Assessment of serve speed (radar) during 15 serves

Second session :

* Clinical testing

  a. Assessment of rotator cuff muscles strength
* Functional tests

  1. Lateral Medecine Ball throw (5 repetitions)
  2. Single arm ball throw (1,5kg)

ELIGIBILITY:
Inclusion Criteria:

* playing tennis at a level of ITN2-4
* being healthy

Ages: 14 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Forty healthy tennis players (aged 14-30) and ITN 2-4 will be recruted in the clubs of the Province of Liege.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Shoulder range of motion | through study completion, an average of 3 months
  Internal/external rotation range of motion assessment
Shoulder strength | through study completion, an average of 3 months
  Internal/external rotators strength measurement
Serve speed | through study completion, an average of 3 months
  Measurement of serve speed with a radar
Upper extremity Y balance test | through study completion, an average of 3 months
  Maximal score in the 3 directions will be retained
Lateral Medicine Ball Throw | through study completion, an average of 3 months
  Measurement of the time to do 5 repetitions
Single Arm ball throw | through study completion, an average of 3 months
  Measurement of the maximal distance reached

CONTACTS AND LOCATIONS:
Locations (1):
- Tennis Club in the Province of Liege, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No